CLINICAL TRIAL: NCT01409265
Title: The Impact of Perceptual Impairment on Social Participation in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: 99-3385B
Record Dates: First submitted 2011-03-17; First posted 2011-08-04 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2014-09

CONDITIONS: Cerebrovascular Accidents
Keywords: stroke rehabilitation; perceptual deficits
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
The perceptual change on stroke patients during the movement recovery and its relationship with social participation still remain unclear. The purposes of this study are: 1) to observe the progression of perception deficit and 2) to understand the relationships among perception deficit and other functional indicators.

A total of 90 stroke patients will be recruited. Each patient will receive three times evaluation, including perception tests, motor function test, daily living ability tests and social leisure participation questionnaires.

DETAILED DESCRIPTION:
According to motor control theory, perception plays an important role in the execution of motion. Although the effect of rehabilitation for motor recovery on stroke patients has been well established, the perceptual change during the movement recovery and its relationship with social participation still remain unclear.

A total of 90 stroke patients will be recruited. Each patient will receive initial evaluation, first follow-up evaluation after four weeks and second follow-up evaluation after five months. The contents include basic clinical screen tests, perception tests, motor function test, daily living ability tests and social leisure participation questionnaires.

The purposes of this study are: 1) to observe the change of the during the experiment and clarify the progression of perception deficit and 2) to understand the relationships among perception deficit and the other functional indicators and determine the impact of perception deficit on activities and participation in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* the age over 40 years old
* the time of onset more than 3 months
* no cognitive dysfunction
* cerebral stroke
* clinical diagnosis of a first or recurrent unilateral stroke

Exclusion Criteria:

* recurrent of the stroke or epilepsy during the intervention
* patients with the neurological or psychical history, for example, alcoholism, drug poisoning or bipolar disorder
* participate in the other interventional study in the same time
* refuse subscribed the informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the rehabilitation department of hospitals
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | Up to 3 years
  The FMA is used to evaluate stroke-related motor impairment, including upper- and lower-extremity movements, sensation, and balance. The whole FMA takes approximately 30 to 40 minutes to administer. The upper-extremity subscale of the FMA contains 33 items to assess motor impairment. Each item is scored on a 3-point ordinal scale (0-cannot perform, 1-performs partially, 2-performs fully and correctly). It is administered 3 times during the study period.

SECONDARY OUTCOMES:
Box and Block Test (BBT) | Up to 3 years
  The BBT is a test of manual dexterity and was originally developed to evaluate the gross manual dexterity of adults with cerebral palsy. A box with a partition directly in the center creating two equal sides is used in the test. Small wooden blocks are placed in one side of the box. The participant is required to use the unaffected had to grasp one block at a time and transport it over the partition and release it into the opposite side. 60 seconds is given to complete the test, and the number of blocks transported to the other side is counted. Then the participant is asked to repeat the same task with the affected hand. The BBT is administered 3 times during the study period.
Modified Ashworth Scale (MAS) | Up to 3 years
  The MAS is a 5-point ordinal scale to evaluate muscle tone of upper-extremity. Higher scores indicate a more severe hypertonia. This measure is administered 3 times during the study period.
Medical Research Council scale (MRC) | Up to 3 years
  The MRC scale assesses muscle power with scores ranging from 0 (no contraction) to 5 (normal power). The muscle strength of shoulder flexors/abductors, elbow flexors/extensors, wrist flexors/extensors, and finger extensors are graded. The MRC is administered 3 times during the study period.
Wolf Motor Function Test (WMFT) | Up to 3 years
  The WMFT is used to assess the upper extremity function. The WMFT consists of 17 tasks, including 15 function tasks and 2 strength tasks. We only used the sum of the 15 functional tasks. The 15 functional tasks are timed (WMFT-TIME) and rated by using a 6-point functional ability scale (WMFT-FAS) where 0 indicates "does not attempt with the involved arm" and 5 represents "arm does participate; movement appears to be normal." The maximum score is 75. Higher scores are indicative of higher functioning levels. The WMFT is administered 3 times during the study period.
Action Research Arm Test (ARAT) | Up to 3 years
  The ARAT is used to evaluate upper extremity function. It consists of 19 items, and tasks are scored on a 4-point scale. A maximum of a total score 57 indicates normal performance. This measure is administered 3 times during the study period.
Nottingham Extended Activities of Daily Living Scale (NEADL) | Up to 3 years
  The NEADL scale is a measure of Instrumental ADL ability, comprising sub-scales for mobility, household ability and leisure activity. The NEADL consists of 22 activity items, scoring on the basis of the required level of assistance. The range of total score is 0-66, and higher score representing better function. This measure is administered 3 times during the study period.
Adelaide Activities Profile (AAP) | Up to 3 years
  The AAP is used to assess life-style activities of the elderly. The AAP asks elderly people to provide responses which reﬂect their performance of 21 activities in a typical three-month period. Each activity is rated using four possible responses, scored 0, 1, 2 or 3 to indicate increasing frequency of activity. It consists of activities in domestic chores, household maintenance, service to others, and social activities. This measure is administered 3 times during the study period.
ABILHAND questionnaire | Up to 3 years
  The ABILHAND questionnaire is a self report assessment that assesses the UE function that consists of 23 bilateral activities in the daily life. Patients were asked to estimate their difficulty in performing each activity.The ABILHAND is a 3-point ordinal scale, which the higher scores mean the more difficulty patients feel. This measure is administered 3 times during the study period.
Motor Activity Log (MAL) | Up to 3 years
  The MAL is a semi-structured interview of patients to assess the amount of use (AOU) and quality of movement (QOM) of the affected upper extremity in 30 important daily activities using a 6-point ordinal scale. Higher scores indicate superior amount and quality of use in affected upper extremity. Each task is scored on a 6-point scale, ranging from 0 to 5. This measure is administered 3 times during the study period.
Stroke Impact Scale Version 3.0 (SIS 3.0) | Up to 3 years
  The SIS 3.0 is a stroke-specific instrument of health-related quality of life and contains 59 items measuring 8 domains. Items are rated on a 5-point Likert scale with lower scores indicate greater difficulty in task completion during the past week. Aggregate scores, ranges from 0 to 100, are generated for each domain. It is administered 3 times during the study period.
Nottingham Leisure Questionnaire (NLQ) | Up to 3 years
  The NLQ was developed to measure such decline in patients with a stroke and to monitor the effects of interventions on leisure. The NLQ lists 37 leisure items and has five possible response categories (very regularly, regularly, occasionally, infrequently, never). Higher scores denote a greater number of activities performed and/or greater frequency of activity. This measure is administered 3 times during the study period.
Leisure Satisfaction Scale (LSS) | Up to 3 years
  The LSS evaluates the extent to which individuals feel that their needs are met through their leisure activities. The LSS included 24 Likert scale items (1=strongly disagree, 5=strongly agree). Categories included psychological, educational, social, relaxational, physiological, and aesthetic effects. A total score for each area and overall LSS score are calculated. This measure is administered 3 times during the study period.
Reintegration to Normal Living Index (RNLI) | Up to 3 years
  The RNLI is an assessment of the quality of life (QOL) of people with disabilities. It includes 11 items. Concepts measured by the RNLI include mobility, self-care, daily activity, recreational activity, and family roles. The 100-point scale used a visual analog scale (VAS) anchored by opposing phrases. Higher scores indicate better QOL. This measure is administered 3 times during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-yi Wu, ScD, Study Director — Department of Occupational Therapy, Chang Gung University
Locations (1):
- Chia-ling Chen, Kwei-Shan, Toayuan County, Taiwan